CLINICAL TRIAL: NCT05857254
Title: What Treatment Adherence for Home Parenteral Nutrition in Patients With Chronic Intestinal Failure ?
Brief Title: Treatment Adherence of Home Parenteral Nutrition in Patients With Chronic Intestinal Failure. (QANPIC)
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/09
Record Dates: First submitted 2023-04-20; First posted 2023-05-12 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Chronic Intestinal Failure
Keywords: Chronic intestinal failure; Treatment adherence
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic intestinal failure patient: Patient with chronic intestinal failure and with home parenteral nutrition treatment stable for at least 3 months and with home parenteral nutrition treatment for at least 6 months.
  Interventions: Other: Patient with chronic intestinal failure

INTERVENTIONS:
Other: Patient with chronic intestinal failure — The negociation component will be assessed during an office visit with the help of forms, by the difference between " ideal " parenteral nutrition prescription proposed by prescriber and the " final " prescription, that the patient ultimately receives at the end of the office visit.
  The compliance component will be assessed by a telephone interview, 8 weeks after the office visit.

SUMMARY:
This observational, cross-sectionnal, multicentric study evaluates treatment adherence of home parenteral nutrition in patients with chronic intestinal failure.

DETAILED DESCRIPTION:
Chronic intestinal failure (CIF) is a chronic disease and its main treatment is home parenteral nutrition. This disease is defined by a small bowel dysfunction preventing absorption of nutrients and water inputs. A " normal " oral diet is then insufficient, and must be supplied by an " artificial " parenteral nutrition. This treatment is administered at home, by a central veinous catheter, with varying volumes and frequencies.

The quality of life of patients treated by home parenteral nutrition is significatively altered .

The constraints linked to this treatment may make it difficult to follow. The patients can be lead to ask their doctor for a relief or a modification of this treatment during office visits, to improve their quality of life.

Poor treatment adherence concerns 25% of patients with chronic disease . It has never been assessed in France in CIF.

The goal of this study is to evaluate the treatment adherence for home parenteral nutrition in two of its components: negotiation during office visits, and compliance at home.

The negociation component will be assessed during an office visit with the help of forms, by the difference between " ideal " parenteral nutrition prescription proposed by prescriber and the " final " prescription, that the patient ultimately receives at the end of the office visit.

The compliance component will be assessed by a telephone interview, 8 weeks after the office visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Diagnosis of CIF (insufficiency of intestinal absorptive, motor or vascular functions that require parenteral nutrition).
* Home parenteral nutrition treatment for at least 6 months.
* With home parenteral nutrition treatment stable for at least 3 months.
* Agreeing to participate in research protocol.

Exclusion Criteria:

* Any condition that does not let a telephone interview (example : deafness, severe neurocognitive impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with chronic intestinal failure
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Difference in the volume of parenteral nutrition | Inclusion visit, 8 weeks
  A 10% (or more) difference between " ideal " and " final " prescriptions (one week's assessment of volume difference in mL) And/or During telephone survey, highlighting a 10% (or more) difference in nutrition received, compared to what is indicated on the prescription (assessment done on the difference in volume in mL over a week).

SECONDARY OUTCOMES:
Patient's compliance | Inclusion visit
  Evaluation of the " perception of patients'compliance " by the coordinating nurse of the nutrition center by an analog visual scale. Analog visual scale is scored from 0 (good compliance) to 10 (poor compliance)
Anxiety and depression symptom | Inclusion visit
  Identification of signs of anxiety and depression symptoms by the HADS form. The anxiety and depression scale consists of 14 questions that assess how subjects feel at the time and generally.
Patient's trust | Inclusion visit
  Evaluation of patient's trust in their specialist physician by the WFPTS form. This scale assesses the patient trust's in their specialist ; it consists in 10 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Florian POULLENOT, MD, Principal Investigator — University Hospital, Bordeaux
Locations (6):
- France (6):
  - CHU de Grenoble, Grenoble
  - CHU Limoges, Limoges
  - Institut régional du cancer Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - Hôpital de l'Archet, Nice
  - CHU Bordeaux, Pessac